CLINICAL TRIAL: NCT05721131
Title: NC Thermometer (Gen 3) ISO 80601-2-56 Validation
Status: Completed | Type: Observational
Sponsor: Natural Cycles (Industry)
Responsible Party: Sponsor
Other Study IDs: 2023001
Record Dates: First submitted 2023-01-31; First posted 2023-02-09 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Febrile Illness; Healthy; Fever
MeSH Terms: conditions — Fever

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (1):
- Temperature measurement: Each subject will have their temperature measured by both the NC° Thermometer (Gen 3) and the reference clinical thermometer.
  Interventions: Device: NC° Thermometer (Gen 3)

INTERVENTIONS:
Device: NC° Thermometer (Gen 3) — The NC° Thermometer (Gen3) is used orally for the intermittent measurement and monitoring of human body temperature. The device can be used by adults and children over the age of 5 years old.

SUMMARY:
The purpose of this clinical validation is to evaluate the the clinical bias, the limits of agreement, and the clinical repeatability of measuring oral temperature using a new thermometer, NC° Thermometer (Gen 3), compared to a reference clinical thermometer.

DETAILED DESCRIPTION:
The purpose of this clinical study is to validate the clinical accuracy of the NC° Thermometer (Gen 3) according to the requirements of ISO 80601-2-56:2017. The NC° Thermometer (Gen 3) (the device under study (DUT)) is a predictive thermometer that operates in adjusted mode. The Welch Allyn oral thermometer (Welch Allyn Spot Vital Signs 420 SureTemp temperature module, Welch Allyn, San Diego, CA) with a measurement accuracy of ± 0.1 °C in monitor mode will be used the reference clinical thermometer (RCT). During the clinical study, subjects will be asked to perform three consecutive oral measurements with the DUT, and one oral measurement with the RCT.

ELIGIBILITY:
Inclusion Criteria:

* They are more than 5 years old
* They have not taken any antipyretic in the preceding 120 minutes
* They have no medical conditions which might impact the clinical accuracy validation results, such as inflammation at the measuring site (the mouth)
* They are not taking medications such as barbiturates, thyroid preparations, antipsychotics, and recent immunizations

Min Age: 5 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Subjects will be asked to participate and enrolled during standard visits to the medical clinic or office location.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2023-04-27 (Actual); Study Completion 2023-04-27 (Actual)

PRIMARY OUTCOMES:
Clinical Bias | Up to 1 hour
  Clinical bias is the mean difference between the output temperatures of the NC° Thermometer (Gen 3) (DUT) and the reference clinical thermometer (RCT) for a specific reference body site (the mouth) when measured from a selected group of subjects. The clinical bias of the DUT defines closeness between the DUT output temperature and that of the RCT.
Limits of agreement | Up to 1 hour
  Dispersion of output temperatures around the clinical bias can be estimated by the standard deviation of the temperature differences between the DUT and the RCT as measured from multiple subjects.
Clinical repeatability | Up to 1 hour
  Clinical repeatability (sometimes called the perceived accuracy) is a measure of the consistency of repeated measurements with identical operating conditions when temperatures are taken within short time intervals from the same measuring site of the same subject by the same operator with the same intermittent clinical thermometer. Clinical repeatability is a pooled standard deviation of triplicate measurements over the population of subjects.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Choice Health Network- Reyes Health Center, Anaheim, California
  - Natural Cycles, New York, New York

IPD SHARING:
Plan to Share IPD: No